CLINICAL TRIAL: NCT07218302
Title: Optimizing an Automated Chatbot to Achieve Efficient, Scalable Treatment for Eating Disorders
Brief Title: Eating Disorder Chatbot Optimization
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: New York University (Other); University of South Carolina (Other)
Responsible Party: Principal Investigator, Ellen E. Fitzsimmons-Craft, Associate Professor of Psychological & Brain Sciences and Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 202505037
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Eating Disorders
Keywords: Eating Disorder Intervention; Eating Pathology; Eating Disorder Symptoms; Digital Mental Health; Chatbot; Optimization Randomized Control Trial; Multiphase Optimization Strategy
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Chatbot targeting weight & shape over-evaluation (WSC) (Experimental): Participant will have access to the chatbot component addressing weight & shape over-evaluation. Participant will receive scheduled targeted practice for the weight & shape over-evaluation component. At any time, participant will have access to initiate practice in assigned study component.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting dietary restraint (DR) (Experimental): Participant will have access to the chatbot component addressing dietary restraint. Participant will receive scheduled targeted practice for the dietary restraint component. At any time, participant will have access to initiate practice in assigned study component.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting emotion dysregulation (ED) (Experimental): Participant will have access to the chatbot component addressing emotion dysregulation. Participant will receive scheduled targeted practice for the emotion dysregulation component. At any time, participant will have access to initiate practice in assigned study component.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting resisting urges to binge (UB) (Experimental): Participant will have access to the chatbot component addressing resisting urges to binge. Participant will receive scheduled targeted practice for the resisting urges to binge component. At any time, participant will have access to initiate practice in assigned study component.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting WSC and DR (Experimental): Participant will have access to the chatbot components addressing weight & shape over-evaluation and dietary restraint. Participant will receive scheduled targeted practice for the weight & shape over-evaluation and dietary restraint components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting WSC and ED (Experimental): Participant will have access to the chatbot components addressing weight & shape over-evaluation and emotion deregulation. Participant will receive scheduled targeted practice for the weight & shape over-evaluation and emotion dysregulation components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting WSC and UB (Experimental): Participant will have access to the chatbot components addressing weight & shape over-evaluation and resisting urges to binge. Participant will receive scheduled targeted practice for the weight & shape over-evaluation and resisting urges to binge components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting DR and ED (Experimental): Participant will have access to the chatbot components addressing dietary restraint and emotion deregulation. Participant will receive scheduled targeted practice for the dietary restraint and emotion dysregulation components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting DR and UB (Experimental): Participant will have access to the chatbot components addressing dietary restraint and resisting urges to binge. Participant will receive scheduled targeted practice for the dietary restraint and resisting urges to binge components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting ED and UB (Experimental): Participant will have access to the chatbot components addressing emotion dysregulation and resisting urges to binge. Participant will receive scheduled targeted practice for the emotion dysregulation and resisting urges to binge components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting ED; UB; and DR (Experimental): Participant will have access to the chatbot components addressing emotion dysregulation, resisting urges to binge, and dietary restraint. Participant will receive scheduled targeted practice for the emotion dysregulation, resisting urges to binge, and dietary restraint components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting ED; UB; and WSC (Experimental): Participant will have access to the chatbot components addressing emotion dysregulation, resisting urges to binge, and weight and shape over-evaluation. Participant will receive scheduled targeted practice for the emotion dysregulation, resisting urges to binge, and weight and shape over-evaluation components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting ED; DR; and WSC (Experimental): Participant will have access to the chatbot components addressing emotion dysregulation, dietary restraint, and weight and shape over-evaluation. Participant will receive scheduled targeted practice for the emotion dysregulation, dietary restraint, and weight and shape over-evaluation components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting UB; DR; and WSC (Experimental): Participant will have access to the chatbot components addressing resisting urges to binge, dietary restraint, and weight and shape over-evaluation. Participant will receive scheduled targeted practice for the resisting urges to binge, emotion dysregulation, dietary restraint and weight, and shape over-evaluation components. At any time, participant will have access to initiate practice in assigned study components
  Interventions: Behavioral: Digital Chatbot Program
- Chatbot targeting UB; DR; ED; and WSC (Experimental): Participant will have access to the chatbot components addressing resisting urges to binge, dietary restraint, emotion dysregulation, and weight and shape over-evaluation. Participant will receive scheduled targeted practice for the resisting urges to binge, emotion dysregulation, dietary restraint, emotion dysregulation, and weight and shape over-evaluation components. At any time, participant will have access to initiate practice in assigned study components.
  Interventions: Behavioral: Digital Chatbot Program
- Referral to seek services (No Intervention): Those randomized to receive all chatbot components "off" will receive a referral to seek services.

INTERVENTIONS:
Behavioral: Digital Chatbot Program — Wysa is a digital rules-based chatbot program platform offering cognitive-behavioral therapy-based guided self-help modules. Participants in an arm with access to Wysa will engage with the digital chatbot program daily for eight weeks.
  Arms: Chatbot targeting DR and ED; Chatbot targeting DR and UB; Chatbot targeting ED and UB; Chatbot targeting ED; DR; and WSC; Chatbot targeting ED; UB; and DR; Chatbot targeting ED; UB; and WSC; Chatbot targeting UB; DR; ED; and WSC; Chatbot targeting UB; DR; and WSC; Chatbot targeting WSC and DR; Chatbot targeting WSC and ED; Chatbot targeting WSC and UB; Chatbot targeting dietary restraint (DR); Chatbot targeting emotion dysregulation (ED); Chatbot targeting resisting urges to binge (UB); Chatbot targeting weight & shape over-evaluation (WSC)

SUMMARY:
The purpose of this study is to optimize an automated digital chatbot intervention for adults with clinical or subclinical eating disorders.

DETAILED DESCRIPTION:
Eating disorders (EDs) are common-affecting an estimated 10% of individuals in their lifetimes-and have disabling consequences being associated with high psychiatric comorbidity, impairment, and mortality. Despite this, less than 20% of individuals with an ED ever receive treatment. When individuals do seek treatment, many are not evidence-based and come with high costs and burden on the healthcare system. One solution to this is a chatbot intervention that is evidence-based, affordable, and accessible for people with EDs. This project will assess four candidate components of a cognitive behavioral therapy (CBT)-based chatbot to determine the optimal chatbot package. CBT is the recommended first-line treatment for EDs, yet there is no research to date on which components are most effective or needed for meaningful change in ED psychopathology. In this study the intervention will be divided into four components targeting: (1) over-evaluation of weight and shape; (2) dietary restraint; (3) emotion dysregulation; and (4) resisting urges to binge. The investigators will recruit 800 adults with a binge/purge-type ED who are not currently in treatment and randomly assign participants to one of 16 experimental conditions (each combination from 1 to all 4 components) or the waitlist-control group. Participants will be assessed on changes in ED psychopathology, ED behavior frequencies, comorbid symptoms (i.e., depression, anxiety), and clinical impairment at 1-, 2-, and 6-months following randomization. An optimized package of these candidate components that is most effective, while remaining efficient, will be identified using multiphase optimization strategy (MOST). The investigators' established relationships with industry and non-profit partners will ensure this optimized package has high potential for scalability and dissemination into the community.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Owns a smartphone
* Speaks English
* US resident
* Screens for a clinical or subclinical eating disorder
* Low suicidality
* Not currently in treatment for an eating disorder
* Does not have a medical condition or take medications that impact appetite/weight
* Not currently pregnant

Exclusion Criteria:

* Below 18 years of age
* Does not own a smartphone
* Does not speak English
* Lives outside the US
* Screens as: at risk for an eating disorder, anorexia nervosa, atypical anorexia nervosa, avoidant/restrictive food intake disorder, or not at risk for an ED
* High suicidality
* In treatment for an eating disorder
* Has a medical condition or takes medication(s) that impact appetite/weight
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
ED psychopathology; ED Examination-Questionnaire (EDE-Q) | 6 months
  The EDE-Q is a 28-item inventory derived from an ED diagnostic interview, which asks self-reported concerns with weight and shape, and engagement in ED behaviors, over the last 28 days. Each item is scored from 0-6, with 0 being "No days" and 6 being "Every day". An average is taken of all items participants respond to for a total global score (with possible scores ranging from 0 to 6), where higher scores indicate greater symptomology.

SECONDARY OUTCOMES:
ED behaviors from the EDE-Q; Muscle Building Subscale from the Eating Pathology Symptoms Inventory (EPSI) | 6 months
  The EDE-Q will also be used to gauge self-reported engagement in ED behaviors. Additionally, the EPSI Muscle Building subscale will be used which is a 5-item questionnaire that asks self-reported frequency of muscle building behaviors and attitudes over the last 28 days. Each item is scored from 0 ("Never") to 4 ("Very Often"). Subscale score is calculated by summing items participants respond to (scores may range from 0 to 20), and higher scores indicate greater symptomology.
Depression; Patient Health Questionnaire (PHQ-9) | 6 months
  The PHQ-9 is a 9-item scale asking about self-reported depressive symptoms and suicidality over the past two weeks. All items are scored from 0 ("Not at all") to 3 ("Nearly every day"). Items participants respond to are summed (possible scores ranging from 0 to 27), and higher scores indicate greater symptomology.
Anxiety; Generalized Anxiety Disorder (GAD-7) | 6 months
  The GAD-7 is a 7-item scale assessing self-reported symptoms of anxiety over the past two weeks. All items are scored from 0 ("Not at all") to 3 ("Nearly every day"). Items participants respond to are summed (possible scores ranging from 0 to 21), and higher scores indicate greater symptomology.
Clinical Impairment; Clinical Impairment Assessment (CIA) | 6 months
  The CIA is a 16-item measure that assesses self-reported impairment, or impact on one's life, resulting from eating, weight, or shape in the last 28 days. All items are scores from 0 ("Not at all") to 3 ("A lot"). Items participants respond to are summed (possible scores ranging from 0 to 48), and higher scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Fitzsimmons-Craft, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and informed consent form
Supporting Information: Study Protocol, ICF